CLINICAL TRIAL: NCT02310074
Title: Study on the Efficacy and Safety of Pulsatile Gonadotropin Releasing Hormone Pump Treatment in Patients With Idiopathic Hypogonadotropic Hypogonadism
Brief Title: Efficacy and Safety of Pulsatile Gonadotropin Releasing Hormone Pump Treatment in Patients With Idiopathic Hypogonadotropic Hypogonadism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, the vice-president of Shanghai Jiao Tong University Affiliated Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ruijin-GnRH pump-002
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2014-12

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism | interventions — Chorionic Gonadotropin; Urofollitropin

ARMS (2):
- Pulsatile Gonadotropin Releasing Hormone (Experimental): Pulsatile Gonadotropin Releasing Hormone: subjects in the GnRH group initiated a regimen of pulsatile GnRH administered subcutaneously via a portable infusion pump for 18 months.
  Interventions: Drug: Pulsatile Gonadotropin Releasing Hormone
- combination gonadotropin therapy (Active Comparator): combined human chorionic gonadotropin (hCG)/urinary Follicle-Stimulating Hormone (uFSH) therapy:HCG treatment was maintained alone for 6 months and then uFSH was added for the next 12 months
  Interventions: Drug: Human chorionic gonadotropin; Drug: Urinary Follicle-Stimulating Hormone

INTERVENTIONS:
Drug: Pulsatile Gonadotropin Releasing Hormone
  Other Names: Pulsatile GnRH pump
  Arms: Pulsatile Gonadotropin Releasing Hormone
Drug: Human chorionic gonadotropin — Human chorionic gonadotropin (hCG)
  Arms: combination gonadotropin therapy
Drug: Urinary Follicle-Stimulating Hormone — Urinary Follicle-Stimulating Hormone (uFSH)
  Arms: combination gonadotropin therapy

SUMMARY:
Idiopathic hypogonadotropic hypogonadism (IHH) is the most common disorders of sex development (DSD).Therapy for IHH includes hormone replacement therapy, gonadotropin therapy and pulsed infusion of gonadotropin releasing hormone (GnRH).In the present study, we compared the different efficacy and safety of pulsatile GnRH pump therapy with combination gonadotropin therapy on fertility and sexual development in male patients with IHH.

DETAILED DESCRIPTION:
Idiopathic hypogonadotropic hypogonadism (IHH) is the most common disorders of sex development (DSD).Therapy for IHH includes hormone replacement therapy, gonadotropin therapy and pulsed infusion of gonadotropin releasing hormone (GnRH).In the present study, we compared the different efficacy and safety of pulsatile GnRH pump therapy with combination gonadotropin therapy on fertility and sexual development in male patients with IHH.

The primary endpoint was the achievement of pregnancy in female partner. Secondary endpoints were time to actual attainment of various sperm thresholds: sperm concentration>0*10^6/ml , >1.0 *10^6/ml and >15 *10^6/ml, respectively.

The clinical and laboratory characteristics including testicular and prostatic volume, Tanner stage for pubic hair and genital, serum hormone levels [especially serum testosterone,luteinizing hormone (LH) , and Follicle-Stimulating Hormone (FSH) levels], sperm concentration per ejaculate, and adverse events at baseline and at the end of treatment were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 16 yr
2. Diagnosed as idiopathic hypogonadotropic hypogonadism with clinical signs or symptoms of hypogonadism
3. Hypogonadal serum testosterone levels (<166ng/dl) in the presence of low or normal gonadotropins
4. Normal levels of other anterior pituitary hormones
5. Normal MRI scans of the hypothalamo-pituitary region
6. Had discontinued any prior treatment (testosterone or gonadotropin therapy) for at least three months before enrollment

Exclusion Criteria:

1. With any significant medical condition (including malignant disease), laboratory abnormality, or psychiatric disorders that will prevent the subject from participating in the study
2. Congenital hypopituitarism
3. Any medical or surgical conditions possibly affecting the experiment result
4. Any clinically significant allergic diseases or allergic to the study drugs
5. Recently drug or alcohol abuse(>35unit/week,1unit=8 g alcohol@1 standard drink@250ml beer@140ml wine@25ml strong alcohol drink like whiskey.)

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pregnancy in the female partner | 18 months

SECONDARY OUTCOMES:
first appearance of sperm (month after treatment) | 18 months
first time with sperm density>1*10^6/ml（month after treatment） | 18 months
first time with sperm density>15*10^6/ml（month after treatment） | 18 months

OTHER OUTCOMES:
testicular volume | 18 months
prostatic volume | 18 months
Tanner stage for pubic hair | 18 months
Tanner stage for genital | 18 months
serum hormone levels | 18 months
  especially serum testosterone, LH, and FSH levels
sperm concentration per ejaculate | 18 months
adverse events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD, PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine

REFERENCES:
- [Derived] Yang YY, Zheng SC, Wang WC, Yang ZW, Shan C, Zhang YW, Qi Y, Chen YH, Gu WQ, Wang WQ, Zhao HY, Liu JM, Sun SY. Osteocalcin Levels in Male Idiopathic Hypogonadotropic Hypogonadism: Relationship With the Testosterone Secretion and Metabolic Profiles. Front Endocrinol (Lausanne). 2019 Oct 11;10:687. doi: 10.3389/fendo.2019.00687. eCollection 2019. PMID 31681165